CLINICAL TRIAL: NCT06162988
Title: A Study to Evaluate 5T4 Expression in Malignant Tumors Using 68Ga-NOTA-H006
Brief Title: PET Imaging of 68Ga-NOTA-H006 in Malignancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YiHui Guan (Other)
Responsible Party: Sponsor-Investigator, YiHui Guan, Professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-777
Record Dates: First submitted 2023-11-19; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Tumor, Solid
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who underwent 68Ga-NOTA-H006 and 18F-FDG PET/CT (Experimental): 68Ga-NOTA-H006, single dose
  Interventions: Drug: 68Ga-NOTA-H006 is injected intravenously with a dose of 1.8 MBq[0.05MCi]/kg.

INTERVENTIONS:
Drug: 68Ga-NOTA-H006 is injected intravenously with a dose of 1.8 MBq[0.05MCi]/kg. — 68Ga-NOTA-H006：PET imaging； 18F-FDG：PET imaging

SUMMARY:
5T4, also known as trophoblast glycoprotein, is an oncofoetal antigen expressing in fetal development and cancer but rarely in adult. The high expression of 5T4 in malignancy was found be associated with poor clinical outcomes in ovarian, gastric and colorectal cancers. Several antibody drug conjugates are currently under development for cancer therapy in preclinic and clinic stages.

Previously, investigators engineered a 5T4-specific biomolecule with nanomolar binding affinity. Radiolabeling with gallium-68 resulted in 68Ga-NOTA-H006 which showed 5T4 expression in a variety of xenograft models. Thus, the aims of current study are to evaluate the distribution and dosimetry of this novel tracer, and to explore the diagnostic values of 68Ga-NOTA-H006 in malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer clinical trial study subjects must meet all of the following criteria:

  1. Age between 18 and 65 years old.
  2. Pancreatic occupancy is found on imaging and combined with clinical judgment as a patient with pancreatic cancer.
  3. Written informed consent signed by the subject or his/her legal guardian or caregiver.
  4. Willingness and ability to cooperate with all programs of the study.

Lung cancer clinical trial study subjects must meet all of the following criteria:

1. Be between the ages of 18 and 65 years old.
2. Patients with CT findings of suspicious space on the lungs with a diameter of more than 1cm who have not undergone surgery.
3. Written informed consent must be signed by the subject or his/her legal guardian or caregiver.
4. Willingness and ability to cooperate with all programs of the study.

Bowel cancer clinical trial study subjects must meet all of the following criteria:

1. Be between the ages of 18 and 65.
2. Have a clear histologic or pathologic diagnosis of colorectal cancer.
3. Written informed consent signed by the subject or legal guardian or caregiver.
4. Willingness and ability to cooperate with all programs of this study.

Exclusion Criteria:

1. Severe hepatic or renal insufficiency;
2. Targeted therapy prior to radiotherapy or PET/CT scan. 5T4 expression in existing lesions assessed by immunohistochemistry using antibody clones.
3. History of serious surgery in the last month.
4. Those who have participated in other clinical trials during the same period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Establishment and optimization of imaging method for 68Ga-NOTA-H006 PET | 90mins from time of injection
  Analyze the standardized uptake value (SUV) of 68Ga-NOTA-H006 on the lesions Compare the SUV with 5T4 expression in pathological specimens

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China